CLINICAL TRIAL: NCT03534518
Title: Body Weight Supported Overground Gait Training to Promote Recovery of Walking Function in Chronic Spinal Cord Injury: a Randomized Clinical Trial
Brief Title: Body Weight Supported Training Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Foundation Wings For Life (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-00811
Record Dates: First submitted 2018-05-07; First posted 2018-05-23 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2023-09

CONDITIONS: Spinal Cord Diseases
MeSH Terms: conditions — Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCI-patients receiving overground training (Active Comparator)
  Interventions: Other: BWS overground training
- SCI-patients receiving treadmill training (Active Comparator)
  Interventions: Other: BWS treadmill training

INTERVENTIONS:
Other: BWS overground training — BWS will be provided with the goal to impose the maximal lower extremity weight bearing load without excessive knee flexion during stance phase and/ or toe dragging during the swing phase. The walking tasks will be roughly divided into different domains like skilled walking, balance, dual tasking, walking speed, walking endurance.
  Arms: SCI-patients receiving overground training
Other: BWS treadmill training — Training will be conducted on a standard treadmill with an overhead BWS system that can provide active BWS. Participants are allowed to hold the rails but weight bearing is not allowed. BWS will be provided with the goal to impose the maximal lower extremity weight bearing load without excessive knee flexion during stance phase and/ or toe dragging during the swing phase. Main walking tasks will be endurance (walking long distances at preferred speed) and speed (walking at maximal possible speed).
  Arms: SCI-patients receiving treadmill training

SUMMARY:
Successful ambulation at home and in the community is the main goal of gait training after incomplete spinal cord injury. Many different treatment approaches have been recommended to achieve this goal. One established intervention to achieve that in a clinical setting is body weight supported (BWS) treadmill training. However, recent studies have suggested that the most optimal gait training should be conducted overground with appropriate support conditions to enable a physiological gait pattern. The training has to be challenging and patients must participate as active as possible.

In addition becoming a functional walker in real world involves a variety of walking skills like walking on uneven surfaces, walking up and down slopes, climbing stairs and avoid obstacles. It has been shown in humans as well as in animals that greater improvements are achieved in walking function if the training is task specific. Thus a constrained task like BWS treadmill training may not be the optimal training intervention to become a functional community walker.

Even greater improvements can be expected if patients feel safe during the overground walking and train at their individual limits. With FLOAT there is now the possibility to conduct a task specific BWS overground gait training in a safe environment. The robotic device allows patients to perform different walking tasks like walking overground, avoiding obstacles, walking on uneven and sloped surfaces, climbing stairs, walking in narrow spaces. A virtual reality setup was integrated into the system that even can simulate specific walking tasks like target oriented walking or walking in crowded environment. Based on the promising results seen in preclinical and clinical research, the investigators assume that unrestricted transparent BWS overground training that allows task specific training of real world walking tasks will induce greater improvements than conventional BWS treadmill training.

The investigators will compare the effect of an intensive 4 weeks unrestricted BWS overground gait training to 4 weeks of intensive BWS treadmill training. Not only functional outcome like walking speed or capacity will be assessed but also detailed kinematics that will help to identify the mechanisms of the underlying improvements in walking function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Chronic spinal cord injury (>6 months)
* Incomplete traumatic or non-traumatic lesion (AIS C, D) above T12
* Able to walk 10m with or without walking devices or physical assistance
* Mini-Mental state examination score ³26 (test will only be performed if cognitive deficits are suspected)

Exclusion Criteria:

* Walking capacity > 500m in 6mWT
* Current orthopaedic problems
* History of cardiac condition
* Epilepsy
* Potential pregnancy (pregnancy test must be conducted before
* Each neurophysiological testing)Pressure sore stage 2 or higher, located where a harness could affect healing
* Premorbid major depression or psychosis
* Unlikely to complete the intervention or return for follow-up
* Participation in another training study
* Body weight > 120kg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | Change from day 0 at day 28 and at day 56-63 (follow-up)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No